CLINICAL TRIAL: NCT00447564
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study of Probuphine in Patients With Opioid Dependence
Brief Title: Safety and Efficacy of Probuphine in the Treatment of Opioid Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Titan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO-805
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2017-06

CONDITIONS: Opioid Dependence
Keywords: opioid dependence; opioid addiction; buprenorphine; methadone; heroin; implant; opioid withdrawal; opioid pain medication; suboxone
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator)
  Interventions: Drug: Probuphine
- Group B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Probuphine — 4 implants
  Arms: Group A
Drug: placebo — 4 implants
  Arms: Group B

SUMMARY:
Buprenorphine (BPN) is an approved treatment for opioid dependence, however, in taking oral tablets, patients experience withdrawal and cravings when the variable BPN levels in the blood are low. Probuphine is an implant placed just beneath the skin that contains BPN. It is designed to provide 6 months of stable BPN blood levels. This study will test the safety and efficacy of Probuphine in the treatment of patients with opioid dependence.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written informed consent prior to the conduct of any study related procedures
* Male or female, 18-65 years of age
* Meet DSM-IV criteria for current opioid dependence
* Females of childbearing potential and fertile males must use a reliable means of contraception

Exclusion Criteria:

* Current diagnosis of Acquired Immune Deficiency Syndrome (AIDS)
* Presence of aspartate aminotransferase (AST) levels ≥ 3 X upper limit of normal and/or alanine aminotransferase (ALT) levels ≥ 3 X upper limit of normal and/or total bilirubin ≥ 1.5 X upper limit of normal and/or creatinine ≥ 1.5 X upper limit of normal
* Received treatment for opioid dependence (e.g., methadone, BPN), within the previous 90 days
* Current diagnosis of chronic pain requiring opioids for treatment
* Candidates for only short term opioid treatment or opioid detoxification therapy
* Pregnant or lactating females
* Previous hypersensitivity or allergy to BPN- or EVA-containing substances or naloxone
* Current use of agents metabolized through CYP 3A4 such as azole antifungals (e.g., ketoconazole), macrolide antibiotics (e.g., erythromycin), and protease inhibitors (e.g., ritonavir, indinavir, and saquinavir)
* Current anti-coagulant therapy (such as warfarin) or an INR > 1.2
* Meet DSM-IV criteria for current dependence on any other psychoactive substances other than opioids or nicotine (e.g., alcohol, sedatives)
* Current use of benzodiazepines other than physician prescribed use
* Significant medical or psychiatric symptoms or dementia which in the opinion of the Investigators would preclude compliance with the protocol, patient safety, adequate cooperation in the study, or obtaining informed consent
* Concurrent medical conditions (such as severe respiratory insufficiency) that may prevent the patient from safely participating in study; and/or any pending legal action that could prohibit participation and/or compliance in study
* Participated in a clinical study within the previous 8 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2006-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The cumulative distribution function (CDF) of the percent of urine samples negative for illicit opioids | weeks 1-16

SECONDARY OUTCOMES:
The cumulative distribution function (CDF) of the percent of urine samples negative for illicit opioids | weeks 17-24
Mean percent urines negative for illicit opioids | weeks 1-16
Mean percent urines negative for illicit opioids | weeks 17-24
Proportion (percent) of study completers | weeks 1-16
Proportion (percent) of study completers | weeks 17-24
Total number of weeks of abstinence | weeks 1-16
Total number of weeks of abstinence | weeks 17-24
Mean maximal period in weeks of continuous abstinence | weeks 1-16
Mean maximal period in weeks of continuous abstinence | weeks 17-24
Mean total score on the SOWS | weeks 1-16
Mean total score on the SOWS | weeks 17-24
Mean total score on the COWS | weeks 1-16
Mean total score on the COWS | weeks 17-24
Mean subjective opioid cravings assessment (VAS) | weeks 1-16
Mean subjective opioid cravings assessment (VAS) | weeks 17-24
Patient-rated Clinical Global Impression | weeks 1-16
Patient-rated Clinical Global Impression | weeks 17-24
Physician-rated Clinical Global Impression | weeks 1-16
Physician-rated Clinical Global Impression | weeks 17-24

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Synergy Clinical Research Center, National City, California
  - North County Clinical Research, Oceanside, California
  - Amit Vijapura, MD and Associates, Jacksonville, Florida
  - Fidelity Clinical Research, Lauderhill, Florida
  - Scientific Clinical Research, Inc, North Miami, Florida
  - Northwest Behavioral Research Center, Roswell, Georgia
  - Behavioral Biology Research Unit, Johns Hopkins Bayview Campus, Baltimore, Maryland
  - Dual Diagnosis Unit, SSTAR: Stanley Street Treatment and Resources, Inc., Fall River, Massachusetts
  - Wayne State University Department of Psychiatry and Behavioral Neurosciences, Detroit, Michigan
  - Psych Care Consultants Research, St Louis, Missouri
  - New York VA Medical Center, NYU School of Medicine, New York, New York
  - Addiction Institute of New York, New York, New York
  - Duke University Medical Center Addictions Program, Durham, North Carolina
  - Pahl Pharmaceutical Research, LLC, Oklahoma City, Oklahoma
  - University of Pennsylvania Treatment Research Center, Philadelphia, Pennsylvania
  - Providence Behavioral Health Services, Everett, Washington
  - Puget Sound Health Care Systems, Seattle, Washington

REFERENCES:
- [Derived] Ling W, Casadonte P, Bigelow G, Kampman KM, Patkar A, Bailey GL, Rosenthal RN, Beebe KL. Buprenorphine implants for treatment of opioid dependence: a randomized controlled trial. JAMA. 2010 Oct 13;304(14):1576-83. doi: 10.1001/jama.2010.1427. PMID 20940383